CLINICAL TRIAL: NCT04049916
Title: The Efficacy and Safety of Pyronaridine-artesunate Combined With Low Dose Primaquine for Preventing Transmission of P. Falciparum Gametocytes in Sub-Saharan Africa
Brief Title: Pyronaridine-artesunate With Low Dose Primaquine for Preventing P. Falciparum Transmission
Acronym: NECTAR1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17507; INV-002098 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2019-07-12; First posted 2019-08-08 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-07

CONDITIONS: Malaria,Falciparum
Keywords: Primaquine; Pyramax; Euartesim; Dihydroartemisinin-piperaquine; Pyronaridine-artesunate
MeSH Terms: conditions — Malaria, Falciparum | interventions — pyronaridine; Artesunate; pyronaridine tetraphosphate, artesunate drug combination; artenimol; piperaquine; Primaquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single blind randomised controlled trial. The treating physician and staff involved with assessing all laboratory outcomes of the study are blinded, but no placebo will be used. The study pharmacist will be unblinded and responsible for randomisation and treatment administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pyronaridine-artesunate (PA) (Active Comparator): Subjects will receive pyronaridine-artesunate (PA) once daily for 3 days.
  Interventions: Drug: Pyronaridine Tetraphosphate/Artesunate
- PA with single low dose primaquine (PQ) (Experimental): Subjects will receive pyronaridine-artesunate (PA) once daily for 3 days, and a low dose of primaquine (PQ) on the first dat of treatment. PQ dose is at the World Health Organization (WHO) recommended dose of 0.25 mg/kg.
  Interventions: Drug: Pyronaridine Tetraphosphate/Artesunate; Drug: Primaquine Diphosphate
- Dihydroartemisinin-piperaquine (DP) (Active Comparator): Subjects will receive dihydroartemisinin-piperaquine (DP) once daily for 3 days.
  Interventions: Drug: Dihydroartemisinin/Piperaquine
- DP with single low dose primaquine (PQ) (Active Comparator): Subjects will receive dihydroartemisinin-piperaquine (DP) once daily for 3 days., and a low dose of primaquine (PQ) on the first dat of treatment. PQ dose is at the World Health Organization (WHO) recommended dose of 0.25 mg/kg.
  Interventions: Drug: Dihydroartemisinin/Piperaquine; Drug: Primaquine Diphosphate

INTERVENTIONS:
Drug: Pyronaridine Tetraphosphate/Artesunate — Adults: Tablets containing 180 mg pyronaridine-tetraphosphate/60mg artesunate (Pyramax, Shin Poong Pharmaceutical Co.), administered according to weight. Children: Granules containing 60 mg pyronaridine-tetraphosphate/20mg artesunate, administered according to weight.
  Other Names: Pyramax
  Arms: PA with single low dose primaquine (PQ); Pyronaridine-artesunate (PA)
Drug: Dihydroartemisinin/Piperaquine — Tablets containing 40 mg dihydroartemisinin/320 mg piperaquine tablets (Eurartesim, Sigma Tau), administered according to weight.
  Other Names: Euartesim
  Arms: DP with single low dose primaquine (PQ); Dihydroartemisinin-piperaquine (DP)
Drug: Primaquine Diphosphate — Extemporaneous preparation of 1mg/mL primaquine phosphate solution, from tablets containing 30mg primaquine (A-PQ 30®, ACE pharmaceuticals, NL) dissolved in 30mL water with a non-interacting fruit-flavoured syrup. Solution will be given at 0.25mg/kg.
  Other Names: Primaquine
  Arms: DP with single low dose primaquine (PQ); PA with single low dose primaquine (PQ)

SUMMARY:
The purpose of this study is to assess the gametocytocidal and transmission reducing activity of pyronaridine-artesunate (PA) and dihydroartemisinin-piperaquine (DP) with and without a single low dose of primaquine (PQ; 0.25mg/kg). Outcome measures will include infectivity at 2 and 7 days after treatment, the duration of infectivity in the artemisinin combination therapy (ACT) only arms, and the production and detectability of histidine rich protein II.

DETAILED DESCRIPTION:
Protocol will be shared on request

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years and ≤ 50 years
* Absence of symptomatic falciparum malaria, defined by fever on enrolment
* Presence of ≥16 gametocytes/µL (i.e. ≥1 gametocytes recorded in the thick film against 500 white blood cells)
* No allergies to study drugs
* Use of antimalarial drugs over the past 7 days (as reported by the participant)
* Hemoglobin ≥ 9.5 g/dL
* Individuals weighing >< 80 kg
* No evidence of severe or chronic disease
* Written, informed consent

Exclusion Criteria:

* Age < 5 years or > 50 years
* Pregnancy
* Previous reaction to study drugs/known allergy to study drugs
* Signs of severe malaria
* Taking drugs which may be metabolized by cytochrome enzyme CYP2D6 (e.g., flecainide, metoprolol, imipramine, amitriptyline, clomipramine)
* Blood transfusion within the last 90 days
* Patients with clinical signs or symptoms of hepatic injury (such as nausea and/or abdominal pain associated with jaundice) or known severe liver disease (i.e. decompensated cirrhosis, Child-Pugh stage B or C).
* Patients with clinical signs or symptoms of renal impairment or known renal impairment
* Family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to prolong the QTc interval such as history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease.
* Taking drugs that are known to influence cardiac function and to prolong QTc interval, such as class IA and III: neuroleptics, antidepressant agents, certain antibiotics including some agents of the following classes - macrolides, fluoroquinolones, imidazole, and triazole antifungal agents, certain non-sedating antihistaminics (terfenadine, astemizole) and cisapride.
* Consent not given

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Change in mosquito infectivity assessed through membrane feeding assays (day 2) | 2 days (day 0 & 2)
  The proportion of mosquitoes infected, assessed through membrane feeding and measured as oocyst prevalence in mosquitoes dissected on day 2 post feed, compared to baseline

SECONDARY OUTCOMES:
Change in mosquito infectivity assessed through membrane feeding assays (day 7) | 2 days (day 0 & 7)
  The proportion of mosquitoes infected, assessed through membrane feeding and measured as oocyst prevalence in mosquitoes dissected on day 7 post feed, compared to baseline
Mosquito infectivity assessed through membrane feeding assays - inter arm | 3 days (day 0, 2 & 7)
  Mosquito infection prevalence and density, assessed through membrane feeding and measured as oocyst prevalence/density in mosquitoes dissected on day 2 and 7 post feed, compared between study arms
Duration of infectivity | 5-10 days (as described)
  Non PQ arms only: Duration of infectivity will be determined from measures of mosquito infection prevalence, assessed through membrane feeding and measured as oocyst prevalence in mosquitoes dissected on day 0, 2, 7, 10 and 14 post treatment, and then weekly until 2 sequential negative feeds or until day 49.
Area under the curve (AUC) of infectivity/time | 5-10 days (as described)
  Non PQ arms only: AUC will be determined from measures of mosquito infection prevalence and density, assessed through membrane feeding and measured as oocyst prevalence/density in mosquitoes dissected on day 0, 2, 7, 10 and 14 post treatment, and then weekly until 2 sequential negative feeds or until day 49.
Haemoglobin level | 11 days
  Haemolysis will be monitored by measuring haemoglobin levels (g/dL) on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Histidine rich protein 2 (HRP2) concentration | 11 days
  Histidine rich protein 2 (HRP2) protein concentration in plasma will be determined in subsequent lab analysis from samples collected on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Histidine rich protein 2 (HRP2) circulation time | 11 days
  Histidine rich protein 2 (HRP2) protein circulation time will be compared between methods of detection
Histidine rich protein 2 (HRP2) area under the curve (AUC) | 11 days
  Histidine rich protein 2 (HRP2) area under the curve (AUC) will be determined from measures of HRP2 concentration
Rapid diagnostic test result | 11 days
  Varied rapid diagnostic tests based on the detection of HRP2 will be used on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment to determine infection prevalence, for comparison between study arms.
Gametocyte density | 11 days
  Gametocyte density (parasites/microlitre) will be measured by microscopy and by molecular methods on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Gametocyte under the curve (AUC) | 11 days
  Gametocyte area under the curve (AUC) will be determined from measures of density.
Gametocyte prevalence | 11 days
  Gametocyte prevalence (parasites/microlitre) will be measured by microscopy and by molecular methods on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Gametocyte circulation time | 11 days
  Gametocyte circulation time (days) will be determined from measures of prevalence.
Gametocyte sex ratio | 11 days
  Gametocyte density will be determined by molecular methods for males and females separately, allowing analysis of sex ratio (proportion of total that is male) on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Asexual parasite density | 11 days
  Asexual parasite density (parasites/microlitre) will be measured by microscopy and by molecular methods on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Asexual parasite area under the curve (AUC) | 11 days
  Asexual parasite area under the curve (AUC) will be determined from measures of density.
Asexual parasite prevalence | 11 days
  Asexual parasite prevalence (parasites/microlitre) will be measured by microscopy and by molecular methods on days 0, 1, 2, 7, 10, 14, 21, 38, 35, 42 and 49 post treatment.
Asexual parasite circulation time | 11 days
  Asexual parasite circulation time (days) will be determined from measures of prevalence.
Parasite genotype | 1 day
  Parasite merozoite surface protein 2 (MSP2) allelic diversity (presence of distinct alleles) will be determined in subsequent lab analysis from whole blood samples collected at baseline.
Histidine rich protein gene deletion | 1 day
  Deletion (presence/absence) of the HRP2/3 genes will be determined from whole blood samples collected at baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- Malaria Research and Training Centre, Bamako, Mali
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Anonymised individual participant data may be shared on a digital repository or upon reasonable request

REFERENCES:
- [Derived] Stone W, Mahamar A, Sanogo K, Sinaba Y, Niambele SM, Sacko A, Keita S, Youssouf A, Diallo M, Soumare HM, Kaur H, Lanke K, Ter Heine R, Bradley J, Issiaka D, Diawara H, Traore SF, Bousema T, Drakeley C, Dicko A. Pyronaridine-artesunate or dihydroartemisinin-piperaquine combined with single low-dose primaquine to prevent Plasmodium falciparum malaria transmission in Ouelessebougou, Mali: a four-arm, single-blind, phase 2/3, randomised trial. Lancet Microbe. 2022 Jan;3(1):e41-e51. doi: 10.1016/S2666-5247(21)00192-0. PMID 35028628